CLINICAL TRIAL: NCT05917795
Title: Prospective Pilot Study for the Evaluation of Endoscopic Sleeve Gastroplasty With Endomina® for the Treatment of Obesity in Kidney Transplant Candidates
Brief Title: Endoscopic Sleeve Gastroplasty With Endomina® for the Treatment of Obesity in Kidney Transplant Candidates
Acronym: ESGiTXKidney
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5764
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-06

CONDITIONS: Obesity, Morbid; End Stage Renal Disease; Kidney Transplantation; Endoscopic Sleeve Gastroplasty
MeSH Terms: conditions — Obesity, Morbid; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- kidney transplant candidates with obesity (BMI > 35 kg/m2) (Experimental): Subjects with an indication to kidney transplantation that are not listed because of a high BMI according to the policy of the transplant Centre (cut-off 35 kg/m2)
  Interventions: Procedure: Endoscopic Sleeve Gastroplasty (ESG)

INTERVENTIONS:
Procedure: Endoscopic Sleeve Gastroplasty (ESG) — ESG will be performed under general anaesthesia with orotracheal intubation. The Endomina® suturing system (EndoTools Therapeutics S.A., Gosselies, Belgium) mounted on a single channel endoscope (GIF-H190/GIF-HQ190; Olympus Medical Systems Corp., Tokyo, Japan) will be used. This system allows to obtain full thickness gastric sutures through the gastric wall of the gastric body, leaving the antrum and the gastric fundus free. The ESG starts with the reduction of the gastric body, suturing from distal to proximal and starting from the notch of the angulus and ending at the level of the fundus. 4-8 full thickness stitches will be placed, with 2 passes per stitch. The final effect of ESG is the creation of a gastric tubule thus reducing the volume of the stomach. After the procedure, the final shape will be evaluated, to examine any gaps that would require additional closure, and to exclude bleedings and/or other complications.

SUMMARY:
The aim of this pilot prospective interventional study is to evaluate the efficacy of endoscopic sleeve gastroplasty (ESG) in allowing obese subjects (≥35 kg/m2) with end stage renal disease who need of kidney transplantation to reduce their BMI below 35 in order to be inserted in the waiting list BMI. The main question[s] it aims to answer are:

Is the procedure effective in reducing BMI to the target level in 12 months? Which is the effect on weight loss, quality of life and obesity-related comorbidities? Participants will undergo ESG as per standard clinical practice and followed up to 12 months before transplantation and for 12 months after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (i.e., age between 18 and 70 years).
* BMI ≥ 35 kg/m²;
* Patients with chronic kidney disease (CKD) G4-G5 (glomerular filtration rate [GFR] <30ml/min/1.73 m2) who are expected to reach end-stage kidney disease (ESKD) at least 6 to 12 months before anticipated dialysis initiation (pre-emptive transplant candidates) or patients already on haemodialysis when medically stable and kidney failure deemed irreversible;
* Patients not listed because of a high BMI according to the policy of the transplant Centre (cut-off 35 kg/m2);
* Signed informed consent.

Exclusion Criteria:

* Patients on peritoneal dialysis
* Upper gastro-intestinal bleeding (gastric or oesophageal) in the previous six months;
* Ongoing or active malignancy during the last 5 years
* Myocardial infarction during the past 6 months or/and heart failure class III or IV according to the New York Heart association's classification;
* Previous stomach, oesophagus or duodenum surgery;
* Technical non-feasibility in the opinion of the endoscopist;
* Clinical signs of active infection;
* Concomitant unstoppable anticoagulant or anti platelet therapy, except for low dose aspirin (≤ 100 mg);
* Active drugs or alcohol abuse;
* Pregnancy, lactation (desire to become pregnant during study duration);
* Enrolment in other clinical studies;
* Contraindication to general anaesthesia;
* Other conditions to exclude the subject in investigators opinion;
* Refusal to sign informed consent. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-09-24 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Kidney transplant list inclusion | 12 months
  number of patients who achieve a BMI < 35 kg/m² within 12 months post-ESG, allowing them to be included in the kidney transplant list

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy